CLINICAL TRIAL: NCT06429228
Title: Comparison of 1 Versus 2 Days Post-Operative Catheterization After Anterior Colporrhaphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Salvatore, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAT_273219
Record Dates: First submitted 2024-01-24; First posted 2024-05-24 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Catheter Related Complication; Anterior Vaginal Wall Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter removal in postoperative day I (Experimental)
  Interventions: Procedure: Catheter removal after surgery
- Catheter removal in postoperative day II (Experimental)
  Interventions: Procedure: Catheter removal after surgery

INTERVENTIONS:
Procedure: Catheter removal after surgery — Removal of catheter placed during the procedure in first or second post-surgical days.

SUMMARY:
Patients who undergo anterior vaginal wall plastic surgery and place the bladder catheter during surgery are selected. The purpose of the study is to evaluate the presence of statistically significant differences in bladder catheter repositioning within 12 hours after bladder catheter removal in the group of patients in whom the bladder catheter is removed on postoperative day I or II.

Secondary outcomes include evaluation of the incidence of urinary tract infections, number of hospitalization days and total hospitalization costs for patients undergoing anterior vaginal wall surgery in patients in whom the bladder catheter is removed on postoperative day I or II.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Patients who are candidates for cystopexy surgery
* Patients who have consented to the signing of the Informed Consent

Exclusion Criteria:

* Micturition dysfunction with preoperative bladder stagnation > 200 cc at pessary evaluation
* History of recurrent cystitis
* Positive preoperative urine culture
* Azotemia > 40 mg/dL or creatininemia > 1 mg/dL
* Not collected signed consent endorsed
* Diabetes mellitus
* Contraindications to transurethral bladder catheterization
* Major protocol violations due to unforeseen intraoperative complications (bladder and/or rectal damage, severe bleeding with need for urinary monitoring)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
differences in bladder catheter repositioning within 12 hours after bladder catheter removal | 12 hours
  After removal of the bladder catheter, on postoperative day I or II, the appearance of urinary urge will be assessed and, in case of spontaneous urination, the quantity of urine will be measured. In the event that after the waiting time of 6 hours an adequate urination stimulus does not arise, we will proceed with an ultrasound evaluation of bladder stagnation (RV) and the application of the department protocol, as follows:
  * if the sum of diuresis and RV is between 500 and 1000 cc, extemporaneous catheterization and re-evaluation after 4 hours are indicated
  * if the sum of diuresis and RV is > 1000cc, positioning of a bladder catheter and maintenance of the same for 5-7 days with subsequent evaluation is indicated.

SECONDARY OUTCOMES:
incidence of urinary tract infections for patients undergoing cystopexy surgery in patients in whom the bladder catheter is removed on postoperative day I or II. | During hospital stay
  Before removing the catheter, a chemical-physical examination will be carried out; if this is positive, urine culture will be carried out. The diagnosis of urinary tract infection will be made with leukocyturia greater than 25 cells per field, positivity for urinary nitrite, presence of at least 20 bacteria per field, bacteriuria and/or more than 100,000 colony forming units associated with at least one of the following signs (fever, dysuria, increased urinary frequency, suprapubic pain, burning on urination or worsening of urinary incontinence). Patients with a positive culture and/or who show symptoms attributable to urinary tract infection will be subjected to antibiotic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No